CLINICAL TRIAL: NCT03204669
Title: Trace Element Repletion Following Severe Burn Injury
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Mette M Berger, Prof, Centre Hospitalier Universitaire Vaudois
Other Study IDs: X21
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Critical Illness; Nutritional Deficiency; Trace Element Deficiency; Burn Injury
Keywords: Copper; Selenium; Zinc; Continuous renal replacement therapy
MeSH Terms: conditions — Critical Illness; Malnutrition; Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Trace elements replacement

SUMMARY:
Major burn patients are characterized by large exudative losses of Cu, Se and Zn. Trace element (TE) repletion has been shown to improve clinical outcome. The study aimed to check if our repletion protocols were achieving normalization of TE plasma concentrations of major burn patients and if the necessity for continuous renal replacement therapy (CRRT) might increase the needs.

DETAILED DESCRIPTION:
Retrospective analysis of prospectively collected data in burn patients requiring intensive care (ICU) between 1999 and 2015. The cohort was divided into 4 groups according to the protocol changes. Period 1 (P1): 1999-2000, P2: 2001-2005, P3: 2006-2010, P4: 2011-2015. Changes consisted mainly in increasing TE repletion doses and duration. Demographic data, daily TE intakes and weekly plasma concentrations were retrieved for the first 21 ICU-days.

ELIGIBILITY:
Inclusion Criteria:

* Burn injury involving ≥20% body surface (TBSA) (i.e. the threshold for intravenous TE repletion prescription)
* At least one TE plasma concentration during the ICU stay

Exclusion Criteria:

* Comfort care
* Admission >24h after burn injury

Ages: 14 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive burns admissions to the ICU, between June 1st, 1999 and December 31st, 2015 in a Swiss quaternary care hospital (Lausanne University Hospital, Centre Hospitalier Universitaire Vaudois).
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 1999-06-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Trace elements plasma concentration | 21 days
  Copper, Selenium and Zinc plasma concentrations, measured by inductively coupled plasma mass spectrometry (ICP-MS). The recommendation was to check them on a weekly basis.

SECONDARY OUTCOMES:
Number of infectious complications | 21 days
  Infectious complications retrieved from the discharge reports, based on microbiological findings and antibiotherapy introduction or rotation. Multiple positive cultures were considered only once when they were related to a unique infectious episode. Concomitant sites of infection, including primary bloodstream infections, were considered as separate episodes of infections. Episodes of infections due to several microorganisms were considered only once. Infections were defined according to the criteria of the Center for Disease Control (CDC), American Burn Association (ABA) and International sepsis forum.
Length of mechanical ventilation | Up to 120 days
  Number of days on the ventilator by the time the patient is discharged from hospital.
Length of stay | Up to 250 days
  Number of days spent in the ICU by the time the patient is discharged from hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- Lausanne University Hospital (Centre Hospitalier Universitaire Vaudois), Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berger MM. Antioxidant micronutrients in major trauma and burns: evidence and practice. Nutr Clin Pract. 2006 Oct;21(5):438-49. doi: 10.1177/0115426506021005438. PMID 16998143
- [Background] Shenkin A. The key role of micronutrients. Clin Nutr. 2006 Feb;25(1):1-13. doi: 10.1016/j.clnu.2005.11.006. Epub 2006 Jan 10. PMID 16376462
- [Background] Berger MM, Baines M, Raffoul W, Benathan M, Chiolero RL, Reeves C, Revelly JP, Cayeux MC, Senechaud I, Shenkin A. Trace element supplementation after major burns modulates antioxidant status and clinical course by way of increased tissue trace element concentrations. Am J Clin Nutr. 2007 May;85(5):1293-300. doi: 10.1093/ajcn/85.5.1293. PMID 17490965
- [Background] Berger MM, Spertini F, Shenkin A, Wardle C, Wiesner L, Schindler C, Chiolero RL. Trace element supplementation modulates pulmonary infection rates after major burns: a double-blind, placebo-controlled trial. Am J Clin Nutr. 1998 Aug;68(2):365-71. doi: 10.1093/ajcn/68.2.365. PMID 9701195
- [Background] Kurmis R, Greenwood J, Aromataris E. Trace Element Supplementation Following Severe Burn Injury: A Systematic Review and Meta-Analysis. J Burn Care Res. 2016 May-Jun;37(3):143-59. doi: 10.1097/BCR.0000000000000259. PMID 26056754